CLINICAL TRIAL: NCT03527888
Title: A Single-Arm, Open-Label, Multicenter Clinical Trial With Anlotinib Hydrochloride Capsule for Primary Malignant Bone Tumors With Recurrence and Distant Metastases
Brief Title: Study of Anlotinib in Patients With Primary Malignant Bone Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-15-II
Record Dates: First submitted 2018-04-18; First posted 2018-05-17 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Neoplasm of Bone
MeSH Terms: conditions — Bone Neoplasms | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib (Other): Anlotinib QD po and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — Anlotinib QD po and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent

SUMMARY:
To evaluate the safety and efficacy of patients with recurrent and metastatic bone tumors.

ELIGIBILITY:
Inclusion Criteria:

1. The patient volunteered to participate in this study and signed an informed consent;
2. Pathological diagnosis of osteosarcoma, chondrosarcoma, source of undifferentiated pleomorphic sarcoma / malignant fibrous histiocytoma, derived bone giant cell tumor of bone or bone primary Ewing's sarcoma / primitive neuroectodermal tumor (PNET) tumor;
3. All patients were failed in chemotherapy (including anthracycline) or intolerance, recurrence or distant metastasis, and at least one measurable lesion (according to RECIST 1.1 criteria);
4. At the age of 14-70, less than 18 year old patients with body surface area to more than 1.5m2;
5. ECOG PS score: 0~1 score (amputation patient's PS score is 0~2), and the expected survival time is over March;
6. The main organs function within 7 days before the treatment, in accordance with the following criteria: the standard of blood routine examination (in 14 days without blood transfusion): The hemoglobin is greater than or equal to 90g/L (by multiple tumor metastasis induced anemia, hemoglobin = 85g/L); The neutrophil absolute value is more than 1.5 * 109/L; Platelet over 80 * 109/L. biochemical examination should comply with the following criteria: The total bilirubin is less than or equal to 1.5 Long ULN; The alanine aminotransferase and aspartate aminotransferase is less than or equal to 2.5ULN, such as liver metastasis, ALT and AST = 5ULN; The serum creatinine or creatinine clearance rate is greater than 1.5ULN 60ml/min; Doppler ultrasound assessment of the lower limit of normal value is more than the left ventricular ejection fraction (50%).
7. Women of childbearing age should use contraceptive measures must be agreed within 6 months in the study period and after the end of the study (such as IUD, pill or condoms); in the study before entering the group within 7 days of serum or urine pregnancy test is negative, and must be for patients with non lactation; men should agree to use contraceptive measures must be 6 months in the research period and the end of the study period after the patients.

Exclusion Criteria:

- Patients with immunodeficiency, including HIV positive or other acquired, congenital immunodeficiency disease, or organ transplant history Hypertension (systolic BP ≥150 mmHg, diastolic BP ≥90 mmHg) still uncontrollable by one medication Hepatitis B virus patients with active replication (DNA> 500 cps / mL), hepatitis C

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Progress free survival (PFS) | through study completion, an average of 6 month
  From random grouping to the objective progression or death of a tumor

SECONDARY OUTCOMES:
Overall Survival (OS) | through study completion, an average of 10 month
  The time in which the group begins to cause death for any reason

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yao, Principal Investigator — Shanghai 6th People's Hospital
Locations (6):
- China (6):
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Shanghai No.6 People's Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of the Air Force Medical University, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan